CLINICAL TRIAL: NCT06041009
Title: Pancreatic Cancer Screening Through the Detection of Elastase-1 Combined With Other Examinations: A Multicenter, Prospective, Diagnostic Clinical Cohort Study.
Brief Title: Pancreatic Cancer Screening Through the Detection of Elastase-1 Combined With Other Examinations
Status: Recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); First Affiliated Hospital of Guangxi Medical University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); LanZhou University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023SDU-QILU-4
Record Dates: First submitted 2023-08-14; First posted 2023-09-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Pancreatic Diseases; Pancreatic Elastase 1; Pancreatic Neuroendocrine Tumor; Pancreatitis; Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Diseases; Adenoma, Islet Cell; Pancreatitis; Pancreatic Neoplasms | interventions — Histocompatibility Testing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and punctured tissue will be collected.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Patients with PDAC
  Interventions: Diagnostic Test: Pancreatic elastase-1 in blood serum
- Individuals at high risk for PDAC
  Interventions: Diagnostic Test: Pancreatic elastase-1 in blood serum
- Group of neuroendocrine neoplasm of pancreas
  Interventions: Diagnostic Test: Pancreatic elastase-1 in blood serum
- Group of solid pseudopapillary tumor of pancreas
  Interventions: Diagnostic Test: Pancreatic elastase-1 in blood serum
- Group of abnormally elevated CA19-9
  Interventions: Diagnostic Test: Pancreatic elastase-1 in blood serum
- Controls without pancreatic disease or elevated CA19-9
  Interventions: Diagnostic Test: Pancreatic elastase-1 in blood serum

INTERVENTIONS:
Diagnostic Test: Pancreatic elastase-1 in blood serum — Serum samples were collected from each patient to detect serum multiomics and pancreatic elastase-1 (PE-1). We examine multiomics in the pancreatic tissue collected from the patient who had undergone surgery or the necessary puncture examination and signed the informed consent form.
  Other Names: Multiomics in blood serum or tissue

SUMMARY:
This is a prospective cohort study. The investigators enroll subjects with pancreatic ductal adenocarcinoma (PDAC), individuals at high risk for PDAC, patients with other pancreatic diseases, patients with CA19-9 elevation and controls without pancreatic disease. This study aims to establish a diagnostic prediction model by using elastase 1, common clinical serological examinations, and imaging examinations including endoscopic ultrasonography (EUS), and to explore the diagnostic ability of the model in the high-risk population of PDAC. Besides, the investigators search for new biomarkers by multi-omics studies of serum and pancreatic tissues to further improve the diagnostic performance of this model. In conclusion, this study seeks a robust diagnostic prediction model to diagnose PDAC, especially early resectable PDAC.

ELIGIBILITY:
Inclusion Criteria:

Case groups (matching any of the following):

1. Patients with pancreatic cancer with recognized diagnostic criteria or conclusions.
2. Patients who are the high-risk group of pancreatic cancer.
3. Patients with solid pseudo papilloma and neuroendocrine tumors of pancreas with recognized diagnostic criteria or conclusions.
4. Patients with other diseases with abnormally elevated CA19-9.

Control group:

(1) Patients without pancreatic disease assessed by laboratory tests and imaging examinations have no CA19-9 elevation.

Exclusion Criteria:

1. Patients who are younger than 18 years of age.
2. Patients with suspected pancreatic malignant lesions but has no confirmed imaging or pathological diagnosis.
3. Patients who have not signed informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pancreatic cancer patients at high risk, patients with pancreatic cancer, benign pancreatic disease, borderline malignant disease, and abnormal elevation of CA199, as well as patients with other diseases without pancreatic disease are included. The Pancreatic cancer patients at high risk are those which are hereditary pancreatic cancer patients at high risk, chronic pancreatitis, new diabetes mellitus, or PCN pancreatic cystic tumor patients.
Sampling Method: Non-Probability Sample
Enrollment: 2100 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
The diagnostic value (sensitivity, specificity, accuracy, and positive and negative predictive values) | 2 years
  The diagnostic value of diagnostic model in diagnosing PDAC, especially early resectable PDAC.

SECONDARY OUTCOMES:
The diagnostic value (sensitivity, specificity, accuracy, and positive and negative predictive values) | 2 years
  The diagnostic value of diagnostic model versus EUS or other imaging examinations combined with diagnostic model in diagnosing PDAC.
The content of elastase 1 | 2 years
  The content of elastase-1 in cystic fluid and serum are measured (units: ng/dl)
The diagnostic value (sensitivity, specificity, accuracy, and positive and negative predictive values) | 2 years
  The ability of diagnostic models, multi-omics novel tumor markers, and common tumor markers to distinguish PDAC, benign pancreatic disease, borderline malignant disease, patients with abnormally elevated CA199, and controls without pancreatic disease.
The diagnostic value (sensitivity, specificity, accuracy, and positive and negative predictive values) | 2 years
  The diagnostic value of the diagnostic model, new tumor markers of multi-omics, and the common tumor markers to distinguish pancreatic tumors of different sites and sizes.

CONTACTS AND LOCATIONS:
Overall Officials: Ning Zhong, MD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Ning Zhong, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No